CLINICAL TRIAL: NCT06793930
Title: The Effects of a Tailored, Optimised, and Person-centred Critical Pathway to Promote Lifestyle Modification in People With Metabolic Syndrome: A Mixed-methods Study
Brief Title: A Tailored, Optimised, and Person-centred Programme to Promote Lifestyle Modification in People With Metabolic Syndrome
Acronym: TOP-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Shinyi, PhD Candidate, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW 24-306; HKUCTR-3030 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2025-01-10; First posted 2025-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome; Primary Prevention of Atherosclerotic Cardiovascular Disease
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Will receive a 12-week tailored, optimised and person-centred programme for sustainable lifestyle modification
  Interventions: Behavioral: A tailored, optimised, and person-centred critical pathway to promote sustainable lifestyle modification
- Control group (Sham Comparator): Will receive an once-off 15-minute structured education
  Interventions: Other: Brief advice

INTERVENTIONS:
Behavioral: A tailored, optimised, and person-centred critical pathway to promote sustainable lifestyle modification — The TOP-S programme is a nurse-led intervention promoting the maintenance of lifestyle modification
  Arms: Intervention group
Other: Brief advice — once-off brief lifestyle advice lasting for 15 minutes
  Arms: Control group

SUMMARY:
This is a mixed-methods study comprising a 2-arm randomised controlled trial and a qualitative study. This study aims to evaluate the effects of a lifestyle modification on the control of metabolic syndrome, with assessments measured at baseline, immediately at the end of the active phase of intervention (12 weeks) and 8 weeks thereafter (20 weeks). It will be conducted in multiple community centres in Hong Kong. Individuals fulfilling the following eligibility criteria will be recruited:

1) Chinese people with metabolic syndrome defined by the 'Harmonising the metabolic syndrome' (HMS) criteria by three or more abnormal findings out of five components (i.e., raised blood pressure, raised triglycerides, lowered HDL, raised fasting blood glucose, and central obesity)[1]; 2) aged ≥18; 3) community-dwelling; 4) independent in daily living, and 5) possessed a digital device with internet connection. Participants will be randomly allocated in a 1:1 ratio to receive the TOP critical pathway (intervention group) or once-off brief lifestyle advice (control group).

Evaluation outcomes will be measured at baseline (T0), 12 weeks (T1) and 20 weeks (T2) thereafter. The outcome assessment includes Health-Promoting Lifestyle Profile-II (HPLP-II), reversal of metabolic syndrome, defining characteristics of metabolic syndrome (body mass index, systolic and diastolic blood pressure, triglycerides, high-density lipoprotein, fasting blood glucose and waist circumference) and the 12-item Short-Form Health Survey version 2 (SF-12v2). Triglycerides, high-density lipoprotein and fasting blood glucose will be measured using a portable point-of-care analyser.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults with metabolic syndrome defined by the 'Harmonising the metabolic syndrome' (HMS) criteria by three or more abnormal findings out of five defining characteristics (i.e., raised blood pressure, raised triglycerides, lowered high-density lipoprotein, raised fasting blood glucose, and central obesity)
2. aged ≥18
3. community-dwelling
4. independent in daily living
5. possessed a digital device with an internet connection

Exclusion Criteria:

1. Has established atherosclerotic cardiovascular diseases (coronary heart disease, cerebrovascular disease and peripheral arterial disease)
2. Has psychiatric diseases
3. Cannot read Chinese
4. Has impaired communication or cognitive function (as indicated by an Abbreviated Mental Test Score of ≤6)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome reversal | From enrollment to the end of the active phase of programme at 12 weeks and 20 weeks
  The reversal of metabolic syndrome will be determined using the Harmonizing the metabolic syndrome criteria. To be classified as the reversal of metabolic syndrome, participants must have ≤2 of the following: (1) a waist circumference of ≥85 cm in men and ≥80 cm in women; (2) triglycerides <1.7mmol/L and/or on drug treatment as an alternate indicator; (3) HDL <1.0 mmol/L in men and <1.3 mmol/L in women and/or on drug treatment as an alternate indicator; (4) systolic blood pressure ≥130 mmHg and/or diastolic blood pressure ≥85 mmHg and/or on antihypertensive drug treatment as an alternate indicator; and (5) fasting blood glucose ≥5.6 mmol/L and/or on drug treatment as an alternate indicator.

SECONDARY OUTCOMES:
Health-promoting behaviours | From enrollment to the end of the active phase of programme at 12 weeks and 20 weeks
  The 52-item HPLP-II (Chinese version) will be used to measure health promoting behaviour. It comprises six subscales measuring health-promoting lifestyle, health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management. Each item of health behaviour is rated according to the frequency that the respondents practice on a four-point Likert Scale, with 1 indicating 'never', 2 indicating 'sometimes', 3 indicating 'often', and 4 indicating 'routinely'. The total score is the mean of all responses to the 52 items, with sub-scale scores representing the mean of all responses to the corresponding items under each subscale. A higher score indicates better reported health promoting behaviours.
Metabolic syndrome components | From enrollment to the end of the active phase of programme at 12 weeks and 20 weeks
  Metabolic syndrome components include systolic and diastolic blood pressure (mmHg), triglycerides (mmol/L), high-density lipoprotein (HDL in mmol/L) , fasting blood glucose(mmol/L), and waist circumference (cm).Systolic and diastolic blood pressure will be measured using a digital automatic blood pressure monitor with an appropriate size cuff. Participants will be asked to relax and sit quietly for 3-5 minutes before the blood pressure measurement. They will be seated with their arm supported at heart level for the measurement. The measurement of waist circumference will be taken at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Capillary blood samples will be taken in the morning after fasting for 12 hours using the finger prick method. A portable point-of-care analyser (CardioChek Plus) will be used to measure circulating HDL, triglycerides, and fasting blood glucose. BMI (kg/m2)will be calculated as weight (kg)/height (m)^2.
Health-related quality of life | From enrollment to the end of the active phase of programme at 12 weeks and 20 weeks
  The 12-item Chinese (HK) SF-12v2 will be used to measure HRQoL. The SF-12v2 consists of eight subscales that form two summary scores, physical summary score and mental summary score, to reflect people's physical and mental health state. The total score ranges from 0 to 100, with a higher score indicating the better health state.
Blood lipid measures | At baseline (T0), immediately at the end of the active intervention phase (12 weeks after baseline)(T1), and 8 weeks thereafter (20 weeks after baseline) (T2).
  A portable point-of-care analyser (CardioChek Plus) will be used to measure circulating cholesterol (total cholesterol, HDL and LDL). Approximately 15uL of capillary blood sample will be collected at each measurement. (The amendment of the study outcome has been approved by the HKU/HA HKW Institutional Review Board)

CONTACTS AND LOCATIONS:
Locations (1):
- Local community centres, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No